CLINICAL TRIAL: NCT03533855
Title: Quality of Image and Performance Diagnoses of the 3D Sequence of Cholangio-pancreatography MRI in Apnea With Compressed Acquisition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3D CP IRM
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Cholangiopancreatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "CS plus FRFSE (Experimental): we perform a classic Fast Relaxation Fast Spin Echo (FRFSE) 3D MRI and add compressed sensing" sequence
  Interventions: Diagnostic Test: CS plus FRFSE

INTERVENTIONS:
Diagnostic Test: CS plus FRFSE — we perform a classic Fast Relaxation Fast Spin Echo (FRFSE) 3D MRI and add compressed sensing" sequence

SUMMARY:
The sequence of 3D CP-IRM, used in current practice in the protocols of bilio-pancreatic imaging, can be thus optimized to reduce acquisition time, thus the artefacts of movement, in particular in 3T. It remains however to estimate if the quality of obtained image is equivalent at least to that of the conventional sequence, without apnea, 3D CP-IRM.

To summarize, the investigators suggest comparing the classic sequence (Fast Relaxation Fast Spin Echo (FRFSE) 3D) already existing with the same sequence to which will be added a technique of CS allowing its acquisition at shortened time(weather), with respiratory trigger on one hand and in apnea on the other hand. For the patient, this study will have for consequence only the addition of 2 sequence MRI, one of the 2 minutes 30 seconds (with respiratory trigger) and other one of the 20 seconds (in apnea).

ELIGIBILITY:
Inclusion Criteria:

* age> 18
* french understanding and speaking patient
* Pancreatic MRI prescription for bilio-pancreatic pathology
* Patient with medical insurance

Exclusion Criteria:

* previous biliary surgery
* MRI contraindication
* Gadolinium recently injected (48 hours)
* Patient couldn't stay on apnea 20 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
image quality scale | Day 1
  Two senior radiologists will analyse the images of MRI with CS sequence

CONTACTS AND LOCATIONS:
Overall Officials: ZINS Marc, MD, Principal Investigator — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France